CLINICAL TRIAL: NCT03068806
Title: Predictive Coding Abnormalities in Psychosis: EEG and fMRI
Brief Title: Brain Imaging, Attention, and Auditory Processing in Schizophrenia
Status: Completed | Type: Observational
Sponsor: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Judith Ford, Research Scientist and Professor of Psychiatry, San Francisco Veterans Affairs Medical Center
Other Study IDs: MH058262
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Electroencephalography; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Schizophrenia: Individuals who have been previously diagnosed with schizophrenia and meet our research criteria for symptoms indicative of schizophrenia within their lifetime.
  Interventions: Diagnostic Test: Electroencephalography (EEG) and Magnetic Resonance Imaging (MRI)
- Healthy Controls: Individuals who have not met criteria for a psychiatric disorder within their lifetime according to our research criteria for symptoms indicative of a psychiatric disorder.
  Interventions: Diagnostic Test: Electroencephalography (EEG) and Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Diagnostic Test: Electroencephalography (EEG) and Magnetic Resonance Imaging (MRI) — The investigators will use these techniques combined with attention tests, memory tests, and clinical interviews to explore connections between these measures and activity in the brain in patients with a diagnosis of schizophrenia and healthy controls.

SUMMARY:
This is a research study designed to examine how the psychiatric illness called schizophrenia affects brain function and thinking abilities such as attention and memory during simple computer-based tasks, and how measures of brain function are related to performance. The investigators do this by looking at brain activity using electroencephalography (EEG) and magnetic resonance imaging (MRI). The investigators compare participants' results to the activity in their brain as well as clinical measures and questionnaires also completed during this study.

DETAILED DESCRIPTION:
* EEG recording: In this procedure, the researcher will assess the participant's brain function while performing simple computer-based tasks. The computer tasks involve presentation of pictures or sounds to which the participant responds by pressing a button. The investigators will also record some of the participant's own speech sounds and play them back to them. The participant will be given clear instructions and a chance to practice before each task. While you are performing these tasks, the investigator will record the weak electrical signals produced by your brain, or "brain waves", using a technique called electroencephalography (EEG). In order to record the participant's EEG, sensors (small plastic discs) will be attached to specific locations on their scalp. The participant's scalp will be gently scrubbed before the sensors are attached. The sensors are held in place on the scalp using a nylon cap that fits snugly on the head. Sensors will also be attached above and below the participant's eyes and will record their eye movements. It will take approximately one hour to attach the sensors. The entire EEG will take approximately 2-3 hours. Before taking part in the EEG session, please make sure to wash hair and scalp. Do not use conditioner or a 2-in-1 shampoo/conditioner. The participant's hair should be dry before arrival. The investigators ask this in order to make the set-up process go more smoothly.

  * During some tasks, participants will feel a vibratory sensation that is produced with an electrical current and it is possible that it may feel like a slight shock. The current is controlled and cannot reach levels that are painful or dangerous. Every participant experiences this sensation differently, so it is important that participants tell the researchers if the sensation becomes uncomfortable to you so the current can be adjusted or the task can be stopped.
  * Participants may be asked to complete additional EEGs for this study, depending on your interest in participating and your availability. All EEG sessions will last approximately 2 hrs.
* MRI: In the fMRI procedure, we will use a magnet to measure blood flow to participants' brains while they do different tasks. Participants will be asked to lie down on a platform that can be slid into the middle of the magnet. A plastic MRI imaging coil will be placed around participants' heads. You will not come into contact with the coil during the experiment. Foam pads will be placed around the participant's head to limit head movement during the experiment. The investigators will then slide you into the magnet. At different points during the experiment, participants will be asked to do the same tasks they did in the training session prior to the scan. During the scan, participants will be asked to either lie still and rest, or do some tasks like tapping their fingers, remembering letters or digits, or viewing images that are designed to activate different parts of the brain. The entire MRI will take approximately two hours.

  * While performing the MRI, participants may be asked to wear a cap that contains multiple EEG sensors applied to your scalp. A removable gel will be used. The EEG measures electrical activity produced by the brain while participants undergo the MRI. Set up for the EEG will take approximately 30 to 60 minutes.
  * Participants may be asked to repeat an MRI session if the data the study team collects is not usable due to data quality issues, or if the participant is unable to stay awake in the magnet during your scan.
* Brief interview session: There will be a series of questions about participants' education, smoking status, and economic background. Participants will also be given a list of words to read to the researcher. If the participant is a patient diagnosed with one of the above-mentioned psychiatric disorders, they will be asked to participate in an additional interview, lasting about one hour, focusing on how they have been feeling recently.
* Behavioral testing: In this part, the participant will use a touch screen computer, mouse and/or paper and pencil to perform certain visual and auditory tests of your mental abilities. Specifically, these tests will assess participants' memory, attention, language, and motor skills. This testing will last approximately one hour. Depending on the participant's preference, this testing can be done on the same day as an EEG or on a different day. The order of the two sessions does not matter, so long as they occur within one week of each other.

Additional Information:

* If information about a participant's mental health is needed from their current or former doctor(s), they will be asked to sign a separate permission form before the researcher can contact their doctor(s).

ELIGIBILITY:
Inclusion Criteria:

* The subject population will include 18 to 75 year old participants of any gender, race, and ethnicity. All subjects will be able to speak and understand English.

Schizophrenia subjects:

1. Patients must be diagnosed with DSM-IV schizophrenia, schizophreniform, or schizoaffective disorder based on a SCID-P interview.

Comparison subjects:

1. Control participants must not have past or present Axis I diagnosis as determined by the SCID-NP.

Exclusion Criteria:

* All subjects:

  1. A hearing deficit greater than 40dB in both ears detected during the hearing test
  2. Substance dependence, as per clinical judgment, in the past 1 year (except caffeine and nicotine)
  3. A history of significant medical/neurological disease such as cardiac, thyroid, renal, hepatic or neurological
  4. History of head injury with loss of consciousness greater than 15 minutes
  5. Any other condition or medication, which in the opinion of the investigator would preclude participation in the study.
  6. Non-English speaking.

Comparison subjects:

1. Any first-degree relative with schizophrenia or bipolar disorder.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with schizophrenia and meet our research criteria of symptoms indicative of a diagnosis of schizophrenia within their lifetime are eligible for this study.
  Healthy controls who have never met criteria for a psychiatric disorder and meet our research criteria will also be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
EEG | Day 1
  Electroencephalography, measures signals from the brain while participants conduct specific tasks that measure memory and attention.
MRI | Day 1
  Magnetic Resonance Imaging, measures activity in, and takes detailed pictures of the brain while participants conduct specific tasks that measure memory and attention.
Memory and Attention tasks | Day 1
  Tasks involve saying words, pressing buttons at specific times, listening, and viewing pictures.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Ford, PhD, Principal Investigator — San Francisco VA Medical Center
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Becsey L, Malamed S, Radnay P, Foldes FF. Reduction of the psychotomimetic and circulatory side-effects of ketamine by droperidol. Anesthesiology. 1972 Nov;37(5):536-42. doi: 10.1097/00000542-197211000-00016. No abstract available. PMID 4562467
- [Background] Bendikov I, Nadri C, Amar S, Panizzutti R, De Miranda J, Wolosker H, Agam G. A CSF and postmortem brain study of D-serine metabolic parameters in schizophrenia. Schizophr Res. 2007 Feb;90(1-3):41-51. doi: 10.1016/j.schres.2006.10.010. Epub 2006 Dec 6. PMID 17156977
- [Background] Broerse A, Crawford TJ, den Boer JA. Parsing cognition in schizophrenia using saccadic eye movements: a selective overview. Neuropsychologia. 2001;39(7):742-56. doi: 10.1016/s0028-3932(00)00155-x. PMID 11311304
- [Background] Clementz BA, McDowell JE, Zisook S. Saccadic system functioning among schizophrenia patients and their first-degree biological relatives. J Abnorm Psychol. 1994 May;103(2):277-87. PMID 8040497
- [Background] Crawford TJ, Sharma T, Puri BK, Murray RM, Berridge DM, Lewis SW. Saccadic eye movements in families multiply affected with schizophrenia: the Maudsley Family Study. Am J Psychiatry. 1998 Dec;155(12):1703-10. doi: 10.1176/ajp.155.12.1703. PMID 9842779
- [Background] Dedovic K, Renwick R, Mahani NK, Engert V, Lupien SJ, Pruessner JC. The Montreal Imaging Stress Task: using functional imaging to investigate the effects of perceiving and processing psychosocial stress in the human brain. J Psychiatry Neurosci. 2005 Sep;30(5):319-25. PMID 16151536
- [Background] Ford JM, Mathalon DH. Corollary discharge dysfunction in schizophrenia: can it explain auditory hallucinations? Int J Psychophysiol. 2005 Nov-Dec;58(2-3):179-89. doi: 10.1016/j.ijpsycho.2005.01.014. Epub 2005 Aug 31. PMID 16137779
- [Background] Ford JM, Mathalon DH, Marsh L, Faustman WO, Harris D, Hoff AL, Beal M, Pfefferbaum A. P300 amplitude is related to clinical state in severely and moderately ill patients with schizophrenia. Biol Psychiatry. 1999 Jul 1;46(1):94-101. doi: 10.1016/s0006-3223(98)00290-x. PMID 10394478
- [Background] Fukushima J, Fukushima K, Morita N, Yamashita I. Further analysis of the control of voluntary saccadic eye movements in schizophrenic patients. Biol Psychiatry. 1990 Dec 1;28(11):943-58. doi: 10.1016/0006-3223(90)90060-f. PMID 2275952
- [Background] Gordon E, Cooper N, Rennie C, Hermens D, Williams LM. Integrative neuroscience: the role of a standardized database. Clin EEG Neurosci. 2005 Apr;36(2):64-75. doi: 10.1177/155005940503600205. PMID 15999901
- [Background] Green MF. What are the functional consequences of neurocognitive deficits in schizophrenia? Am J Psychiatry. 1996 Mar;153(3):321-30. doi: 10.1176/ajp.153.3.321. PMID 8610818
- [Background] Hashimoto K, Engberg G, Shimizu E, Nordin C, Lindstrom LH, Iyo M. Reduced D-serine to total serine ratio in the cerebrospinal fluid of drug naive schizophrenic patients. Prog Neuropsychopharmacol Biol Psychiatry. 2005 Jun;29(5):767-9. doi: 10.1016/j.pnpbp.2005.04.023. PMID 15939521
- [Background] Hashimoto K, Fukushima T, Shimizu E, Komatsu N, Watanabe H, Shinoda N, Nakazato M, Kumakiri C, Okada S, Hasegawa H, Imai K, Iyo M. Decreased serum levels of D-serine in patients with schizophrenia: evidence in support of the N-methyl-D-aspartate receptor hypofunction hypothesis of schizophrenia. Arch Gen Psychiatry. 2003 Jun;60(6):572-6. doi: 10.1001/archpsyc.60.6.572. PMID 12796220
- [Background] Jaeger J, Berns SM, Czobor P. The multidimensional scale of independent functioning: a new instrument for measuring functional disability in psychiatric populations. Schizophr Bull. 2003;29(1):153-68. doi: 10.1093/oxfordjournals.schbul.a006987. PMID 12908671
- [Background] Katsanis J, Kortenkamp S, Iacono WG, Grove WM. Antisaccade performance in patients with schizophrenia and affective disorder. J Abnorm Psychol. 1997 Aug;106(3):468-72. doi: 10.1037//0021-843x.106.3.468. PMID 9241948
- [Background] Krystal JH, D'Souza DC, Mathalon D, Perry E, Belger A, Hoffman R. NMDA receptor antagonist effects, cortical glutamatergic function, and schizophrenia: toward a paradigm shift in medication development. Psychopharmacology (Berl). 2003 Sep;169(3-4):215-33. doi: 10.1007/s00213-003-1582-z. Epub 2003 Sep 2. PMID 12955285
- [Background] Light GA, Hsu JL, Hsieh MH, Meyer-Gomes K, Sprock J, Swerdlow NR, Braff DL. Gamma band oscillations reveal neural network cortical coherence dysfunction in schizophrenia patients. Biol Psychiatry. 2006 Dec 1;60(11):1231-40. doi: 10.1016/j.biopsych.2006.03.055. Epub 2006 Aug 7. PMID 16893524
- [Background] Kwon JS, O'Donnell BF, Wallenstein GV, Greene RW, Hirayasu Y, Nestor PG, Hasselmo ME, Potts GF, Shenton ME, McCarley RW. Gamma frequency-range abnormalities to auditory stimulation in schizophrenia. Arch Gen Psychiatry. 1999 Nov;56(11):1001-5. doi: 10.1001/archpsyc.56.11.1001. PMID 10565499
- [Background] Malhotra AK, Pinals DA, Weingartner H, Sirocco K, Missar CD, Pickar D, Breier A. NMDA receptor function and human cognition: the effects of ketamine in healthy volunteers. Neuropsychopharmacology. 1996 May;14(5):301-7. doi: 10.1016/0893-133X(95)00137-3. PMID 8703299
- [Background] Mathalon DH, Ford JM. The long and the short of it: influence of interstimulus interval on auditory P300 abnormalities in schizophrenia. Clin Electroencephalogr. 2002 Jul;33(3):125-35. doi: 10.1177/155005940203300309. PMID 12192662
- [Background] McDowell JE, Clementz BA. The effect of fixation condition manipulations on antisaccade performance in schizophrenia: studies of diagnostic specificity. Exp Brain Res. 1997 Jun;115(2):333-44. doi: 10.1007/pl00005702. PMID 9224861
- [Background] McDowell JE, Myles-Worsley M, Coon H, Byerley W, Clementz BA. Measuring liability for schizophrenia using optimized antisaccade stimulus parameters. Psychophysiology. 1999 Jan;36(1):138-41. doi: 10.1017/s0048577299980836. PMID 10098389
- [Background] Oranje B, van Berckel BN, Kemner C, van Ree JM, Kahn RS, Verbaten MN. The effects of a sub-anaesthetic dose of ketamine on human selective attention. Neuropsychopharmacology. 2000 Mar;22(3):293-302. doi: 10.1016/S0893-133X(99)00118-9. PMID 10693157
- [Background] Paul RH, Lawrence J, Williams LM, Richard CC, Cooper N, Gordon E. Preliminary validity of "integneuro": a new computerized battery of neurocognitive tests. Int J Neurosci. 2005 Nov;115(11):1549-67. doi: 10.1080/00207450590957890. PMID 16223701
- [Background] Ross RG, Harris JG, Olincy A, Radant A, Adler LE, Freedman R. Familial transmission of two independent saccadic abnormalities in schizophrenia. Schizophr Res. 1998 Feb 27;30(1):59-70. doi: 10.1016/s0920-9964(97)00133-3. PMID 9542789
- [Background] Sereno AB, Holzman PS. Antisaccades and smooth pursuit eye movements in schizophrenia. Biol Psychiatry. 1995 Mar 15;37(6):394-401. doi: 10.1016/0006-3223(94)00127-O. PMID 7772648
- [Background] Spencer KM, Nestor PG, Niznikiewicz MA, Salisbury DF, Shenton ME, McCarley RW. Abnormal neural synchrony in schizophrenia. J Neurosci. 2003 Aug 13;23(19):7407-11. doi: 10.1523/JNEUROSCI.23-19-07407.2003. PMID 12917376
- [Background] Thaker GK, Ross DE, Cassady SL, Adami HM, Medoff DR, Sherr J. Saccadic eye movement abnormalities in relatives of patients with schizophrenia. Schizophr Res. 2000 Oct 27;45(3):235-44. doi: 10.1016/s0920-9964(99)00193-0. PMID 11042441
- [Background] Tsai G, Coyle JT. Glutamatergic mechanisms in schizophrenia. Annu Rev Pharmacol Toxicol. 2002;42:165-79. doi: 10.1146/annurev.pharmtox.42.082701.160735. PMID 11807169
- [Background] Umbricht D, Koller R, Vollenweider FX, Schmid L. Mismatch negativity predicts psychotic experiences induced by NMDA receptor antagonist in healthy volunteers. Biol Psychiatry. 2002 Mar 1;51(5):400-6. doi: 10.1016/s0006-3223(01)01242-2. PMID 11904134
- [Background] Umbricht D, Schmid L, Koller R, Vollenweider FX, Hell D, Javitt DC. Ketamine-induced deficits in auditory and visual context-dependent processing in healthy volunteers: implications for models of cognitive deficits in schizophrenia. Arch Gen Psychiatry. 2000 Dec;57(12):1139-47. doi: 10.1001/archpsyc.57.12.1139. PMID 11115327
- [Background] Yamada K, Ohnishi T, Hashimoto K, Ohba H, Iwayama-Shigeno Y, Toyoshima M, Okuno A, Takao H, Toyota T, Minabe Y, Nakamura K, Shimizu E, Itokawa M, Mori N, Iyo M, Yoshikawa T. Identification of multiple serine racemase (SRR) mRNA isoforms and genetic analyses of SRR and DAO in schizophrenia and D-serine levels. Biol Psychiatry. 2005 Jun 15;57(12):1493-503. doi: 10.1016/j.biopsych.2005.03.018. PMID 15953485
- [Result] Kort NS, Ford JM, Roach BJ, Gunduz-Bruce H, Krystal JH, Jaeger J, Reinhart RM, Mathalon DH. Role of N-Methyl-D-Aspartate Receptors in Action-Based Predictive Coding Deficits in Schizophrenia. Biol Psychiatry. 2017 Mar 15;81(6):514-524. doi: 10.1016/j.biopsych.2016.06.019. Epub 2016 Jul 1. PMID 27647218
- [Result] Ford JM, Roach BJ, Palzes VA, Mathalon DH. Using concurrent EEG and fMRI to probe the state of the brain in schizophrenia. Neuroimage Clin. 2016 Aug 10;12:429-41. doi: 10.1016/j.nicl.2016.08.009. eCollection 2016. PMID 27622140
- [Result] Mifsud NG, Oestreich LK, Jack BN, Ford JM, Roach BJ, Mathalon DH, Whitford TJ. Self-initiated actions result in suppressed auditory but amplified visual evoked components in healthy participants. Psychophysiology. 2016 May;53(5):723-32. doi: 10.1111/psyp.12605. Epub 2016 Jan 11. PMID 26751981
- [Result] Oestreich LK, Mifsud NG, Ford JM, Roach BJ, Mathalon DH, Whitford TJ. Subnormal sensory attenuation to self-generated speech in schizotypy: Electrophysiological evidence for a 'continuum of psychosis'. Int J Psychophysiol. 2015 Aug;97(2):131-8. doi: 10.1016/j.ijpsycho.2015.05.014. Epub 2015 May 28. PMID 26027781
- [Result] Wynn JK, Jimenez AM, Roach BJ, Korb A, Lee J, Horan WP, Ford JM, Green MF. Impaired target detection in schizophrenia and the ventral attentional network: Findings from a joint event-related potential-functional MRI analysis. Neuroimage Clin. 2015 Jul 31;9:95-102. doi: 10.1016/j.nicl.2015.07.004. eCollection 2015. PMID 26448909
- [Result] Ford JM. Studying auditory verbal hallucinations using the RDoC framework. Psychophysiology. 2016 Mar;53(3):298-304. doi: 10.1111/psyp.12457. PMID 26877116
- [Result] Mathalon DH, Sohal VS. Neural Oscillations and Synchrony in Brain Dysfunction and Neuropsychiatric Disorders: It's About Time. JAMA Psychiatry. 2015 Aug;72(8):840-4. doi: 10.1001/jamapsychiatry.2015.0483. PMID 26039190
- [Result] Wang J, Mathalon DH, Roach BJ, Reilly J, Keedy SK, Sweeney JA, Ford JM. Action planning and predictive coding when speaking. Neuroimage. 2014 May 1;91:91-8. doi: 10.1016/j.neuroimage.2014.01.003. Epub 2014 Jan 11. PMID 24423729
- [Result] Ford JM, Palzes VA, Roach BJ, Potkin SG, van Erp TG, Turner JA, Mueller BA, Calhoun VD, Voyvodic J, Belger A, Bustillo J, Vaidya JG, Preda A, McEwen SC; Functional Imaging Biomedical Informatics Research Network; Mathalon DH. Visual hallucinations are associated with hyperconnectivity between the amygdala and visual cortex in people with a diagnosis of schizophrenia. Schizophr Bull. 2015 Jan;41(1):223-32. doi: 10.1093/schbul/sbu031. Epub 2014 Mar 11. PMID 24619536